CLINICAL TRIAL: NCT03339453
Title: Comparison of Glucagon Administered by Either the Nasal (LY900018) or Intra-muscular (GlucaGen®) Routes in Adult Patients With Type 1 Diabetes Mellitus During Controlled Insulin-Induced Hypoglycemia
Brief Title: A Study of Nasal Glucagon in Participants With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 16547; I8R-MC-IGBI (Other: Eli Lilly and Company); 2017-000249-33 (EudraCT Number)
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Results first posted 2019-09-23 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2018-01

CONDITIONS: Hypoglycemia; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Hypoglycemia; Diabetes Mellitus, Type 1 | interventions — Glucagon-Like Peptide 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nasal Glucagon (Experimental): Single dose of Nasal Glucagon.
  Interventions: Drug: Nasal Glucagon
- Intramuscular Glucagon (Active Comparator): Single intramuscular (IM) dose of Glucagon.
  Interventions: Drug: Intramuscular Glucagon

INTERVENTIONS:
Drug: Nasal Glucagon — Administered nasally
  Other Names: LY900018
  Arms: Nasal Glucagon
Drug: Intramuscular Glucagon — Administered IM
  Other Names: GlucaGen®
  Arms: Intramuscular Glucagon

SUMMARY:
The purpose of this study is to compare a needle-free treatment of hypoglycemia with nasal glucagon (study drug) to a marketed glucagon administered by the intramuscular (IM) route, in participants with type 1 diabetes mellitus (T1DM).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 1 Diabetes Mellitus (T1DM) for at least 2 years and receiving daily insulin since the time of diagnosis

Exclusion Criteria:

* Have a history of hypersensitivity to glucagon or any related products or severe hypersensitivity reactions (such as angioedema) to any drugs
* Have a history of pheochromocytoma (that is, adrenal gland tumor) or insulinoma
* Occurrence of an episode of severe hypoglycemia (defined as requiring the assistance of another person in the 1 month prior to enrolling in the study)
* Have a history of epilepsy or seizure disorder
* Are women who are pregnant or lactating
* Have, except for the current regimen of insulin therapy and concomitant medication, regular use of or intended use of any over-the-counter or prescription medications or nutritional supplements that treat hyperglycemia or insulin resistance or that promote weight loss within 14 days before dosing
* Daily use of systemic beta-blocker, indomethacin, warfarin or anticholinergic drugs
* Require daily insulin treatment greater than (>)1.5 unit/kilograms (U/kg)/body weight

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2017-12-17 (Actual); Study Completion 2018-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- Germany (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Mainz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Neuss

REFERENCES:
- [Derived] Seaquist E, Gimenez M, Yan Y, Matsuhisa M, Kao CY, Wadwa RP, Nagai Y, Khunti K. Nasal Glucagon Reverses Insulin-induced Hypoglycemia With Less Rebound Hyperglycemia: Pooled Analysis of Clinical Trials. J Endocr Soc. 2024 Feb 26;8(4):bvae034. doi: 10.1210/jendso/bvae034. eCollection 2024 Feb 19. PMID 38444629
- [Derived] Suico JG, Hovelmann U, Zhang S, Shen T, Bergman B, Sherr J, Zijlstra E, Frier BM, Plum-Morschel L. Glucagon Administration by Nasal and Intramuscular Routes in Adults With Type 1 Diabetes During Insulin-Induced Hypoglycaemia: A Randomised, Open-Label, Crossover Study. Diabetes Ther. 2020 Jul;11(7):1591-1603. doi: 10.1007/s13300-020-00845-7. Epub 2020 Jun 8. PMID 32514794

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In each period, either 3 milligram (mg) nasal glucagon (NG) or 1 mg intramuscular (IM) Glucagon was administered.
  After a wash-out period of at least 1 day (24 hours) from the first period (first visit), participants crossed over to the alternate glucagon treatment in period 2 (second visit).
Groups:
- NG 1st/IM Glucagon 2nd: Participants received 3 mg of NG at the first treatment visit followed by 1 mg of IM glucagon at the second treatment visit.
- IM Glucagon 1st/NG 2nd: Participants received 1 mg of IM glucagon at the first treatment visit followed by 3 mg of NG at the second treatment visit.
Period: First Visit of Glucagon Treatment
Arm/Group | NG 1st/IM Glucagon 2nd | IM Glucagon 1st/NG 2nd
Started | 35 | 35
Received at Least 1 Dose of Study Drug | 35 | 35
Completed | 35 | 34
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Second Visit for Alternate Glucagon
Arm/Group | NG 1st/IM Glucagon 2nd | IM Glucagon 1st/NG 2nd
Started | 35 | 34
Completed (Completed both inpatient study visits.) | 35 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Glucagon: All enrolled participants who received either 3 mg NG or 1 mg IM Glucagon.
Arm/Group | Glucagon
Number analyzed (Participants) | 70
Age, Continuous [Median (Standard Deviation); unit: years] | 41.7 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 70
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 70
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Germany | 70
Weight [Mean (Standard Deviation); unit: Kilogram (kg)] | 78.79 (13.28)
Height [Mean (Standard Deviation); unit: Centimeter (cm)] | 175.21 (8.43)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m2)] | 25.53 (2.97)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Treatment Success During Controlled Insulin-Induced Hypoglycemia
Description: Treatment success is defined as an increase in plasma glucose to greater than or equal to (≥) 70 milligrams per deciliter (mg/dL) or an increase of ≥20 mg/dL from plasma glucose nadir, without receiving additional actions to increase the plasma glucose concentration. Nadir is defined as the minimum plasma glucose concentration at the time of or within 10 minutes following glucagon administration.
Time Frame: Pre-dose up to 30 minutes post each glucagon administration
Population: All participants who completed both treatment visits with evaluable data.
Measure: Count of Participants; unit: Participants
Groups:
- Nasal Glucagon (NG): Dose of 3 mg nasal glucagon.
- IM Glucagon: Dose of 1 mg IM glucagon.
Arm/Group | Nasal Glucagon (NG) | IM Glucagon
Number analyzed (Participants) | 66 | 66
Participants | 66 | 66
Statistical Analysis 1: Comparison: Nasal Glucagon (NG) vs IM Glucagon; Test type: Non-Inferiority — 95% Confidence Interval of the treatment differences in treatment success rate; Risk Difference (RD) = 0.0, 95% CI 2-sided [-1.52 to 1.52]

2. Secondary Outcome: Pharmacodynamics (PD): Change From Baseline in Maximal Blood Glucose (BGmax)
Time Frame: Pre-dose; 5, 10, 15, 20, 25, 30, 40, 50, 60, and 90 minutes after glucagon administration
Population: All enrolled participants who received at least 1 dose of the study drug with evaluable PD data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligrams per deciliter (mg/dL)
Arm/Group | Nasal Glucagon (NG) | IM Glucagon
Number analyzed (Participants) | 68 | 69
Milligrams per deciliter (mg/dL) | 132 (36) | 161 (29)

3. Secondary Outcome: PD: Time to Maximum Concentration (Tmax) of Baseline-Adjusted Glucose
Time Frame: Pre-dose; 5, 10, 15, 20, 25, 30, 40, 50, 60, and 90 minutes after glucagon administration
Population: All enrolled participants who received at least 1 dose of the study drug with evaluable PD data.
Measure: Median (Full Range); unit: Hour (hr)
Arm/Group | Nasal Glucagon (NG) | IM Glucagon
Number analyzed (Participants) | 68 | 69
Hour (hr) | 1.00 [0.42 to 1.50] | 1.50 [0.83 to 1.50]

4. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time Zero to Tlast (AUC[0-tlast]) of Baseline Adjusted Glucagon
Time Frame: Pre-dose; 5, 10, 15, 20, 25, 30, 40, 50, 60, 90, 120, and 240 minutes after glucagon administration
Population: All enrolled participants who received at least 1 dose of the study drug with evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram*hour per millilitre (pg*hr/mL)
Arm/Group | Nasal Glucagon (NG) | IM Glucagon
Number analyzed (Participants) | 63 | 66
picogram*hour per millilitre (pg*hr/mL) | 2740 (68) | 3320 (40)

5. Secondary Outcome: PK: Maximum Change From Baseline Concentration (Cmax) of Glucagon
Time Frame: Pre-dose; 5, 10, 15, 20, 25, 30, 40, 50, 60, 90, 120, and 240 minutes after glucagon administration
Population: All enrolled participants who received at least 1 dose of the study drug with evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picograms per millilitre (pg/mL)
Arm/Group | Nasal Glucagon (NG) | IM Glucagon
Number analyzed (Participants) | 63 | 66
picograms per millilitre (pg/mL) | 6130 (74) | 3750 (44)

6. Secondary Outcome: PK: Time to Maximum Concentration (Tmax) of Baseline Adjusted Glucagon
Time Frame: Pre-dose; 5, 10, 15, 20, 25, 30, 40, 50, 60, 90, 120, and 240 minutes after glucagon administration
Population: All enrolled participants who received at least 1 dose of the study drug with evaluable PK data.
Measure: Median (Full Range); unit: Hour (hr)
Arm/Group | Nasal Glucagon (NG) | IM Glucagon
Number analyzed (Participants) | 63 | 66
Hour (hr) | 0.25 [0.17 to 0.50] | 0.25 [0.08 to 0.50]

ADVERSE EVENTS:
Time Frame: First dose of study drug (Day 1) until post-study completion (Day 30).
Groups:
- Intramuscular (IM) Glucagon: Dose of 1 mg intramuscular glucagon.
Arm/Group | Nasal Glucagon (NG) | Intramuscular (IM) Glucagon
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/69
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/69
Other Adverse Events (participants affected / at risk) | 34/70 | 35/69
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nasal Glucagon (NG) (N=70) | Intramuscular (IM) Glucagon (N=69)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Ocular discomfort (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 22 (22) | 29 (29)
Vomiting (Gastrointestinal disorders) | 10 (10) | 12 (12)
Nasopharyngitis (Infections and infestations) | 4 (4) | 2 (2)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 11 (13) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-10-12): https://cdn.clinicaltrials.gov/large-docs/53/NCT03339453/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-22): https://cdn.clinicaltrials.gov/large-docs/53/NCT03339453/SAP_001.pdf